CLINICAL TRIAL: NCT00315198
Title: A Randomized Trial Comparing Near Versus Distance Activities While Patching for Amblyopia in Children 3 to <7 Years Old
Brief Title: Trial Comparing Near Versus Distance Activities While Patching for Amblyopia in Children 3 to <7 Years Old
Acronym: ATS6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Roy W. Beck, M.D., Ph.D., Executive Director, Jaeb Center for Health Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-114; 2U10EY011751 (NIH); 5U10EY011751 (NIH)
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2009-05

CONDITIONS: Amblyopia
Keywords: amblyopia; patching; visual activities
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Near activities (Active Comparator): 2 hours of daily patching combined with near visual activities while patching
  Interventions: Device: Eye Patch; Procedure: Near activities
- Distance activities (Active Comparator): 2 hours of daily patching combined with distance visual activities while patching
  Interventions: Device: Eye Patch; Procedure: Distance activities

INTERVENTIONS:
Device: Eye Patch — 2 hours daily patching
  Other Names: Coverlet, 3M Opticlude, Ortopad®
Procedure: Near activities — near visual activities while patching
  Arms: Near activities
Procedure: Distance activities — distance visual activities while patching
  Arms: Distance activities

SUMMARY:
Ths purpose of this study is to determine whether "near" activities enhance the effect of patching on visual acuity improvement in strabismic and anisometropic amblyopia when compared with "distance" activities in the treatment of moderate amblyopia and severe amblyopia in children 3 to <7 years old.

DETAILED DESCRIPTION:
The value of "near visual activities" while patching for amblyopia is controversial. Some pediatric eye care providers currently recommend that the child perform near visual tasks while wearing a patch over the sound eye, while other pediatric eye care providers do not prescribe any specific visual tasks to be performed while the patch is worn.

In previous randomized studies of patching doses for amblyopia conducted by the Pediatric Eye Disease Investigator Group, near visual activities were incorporated into the prescribed treatment regimes. Although different doses of patching, combined with near visual activities, were successful in improving visual acuity in most children, it is unclear whether concurrent near visual activities enhanced the effect of patching.

This study is designed as an efficacy study, making effort to maximize adherence to treatment group assignments.

The study has been designed as a simple trial that, other than the type of amblyopia therapy being determined through the randomization process, approximates standard clinical practice. The two treatment regimens for the 17 week treatment period are: 1) 2 hours of daily patching combined with near visual activities while patching and 2)2 hours of daily patching combined with distance visual activities while patching.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 3 to less than 7 years old with amblyopia due to strabismus, anisometropia, or both.
* Visual acuity in the amblyopic eye must be between 20/40 and 20/400 inclusive, visual acuity in the sound eye 20/40 or better and inter-eye acuity difference > 3 logMAR lines.
* Spectacles, if needed, must be worn for at least 16 weeks or until visual acuity documented to be stable.

Exclusion Criteria:

* Prior amblyopia treatment other than spectacles in the past month.
* More than one month of amblyopia treatment in the past 6 months.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 425 (Actual)
Dates: Start 2005-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 8 weeks

SECONDARY OUTCOMES:
Visual acuity | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Don Lyon, O.D., Study Chair — Indiana University; Jonathan M. Holmes, M.D., Study Chair — Mayo Clinic Department of Ophthalmology
Locations (2):
- United States (2):
  - Indiana University School of Optometry, Bloomington, Indiana
  - Mayo Clinic Department of Ophthalmology, Rochester, Minnesota

REFERENCES:
- [Result] Pediatric Eye Disease Investigator Group. A randomized trial of near versus distance activities while patching for amblyopia in children aged 3 to less than 7 years. Ophthalmology. 2008 Nov;115(11):2071-8. doi: 10.1016/j.ophtha.2008.06.031. Epub 2008 Sep 11. PMID 18789533
- [Derived] Wallace DK, Lazar EL, Melia M, Birch EE, Holmes JM, Hopkins KB, Kraker RT, Kulp MT, Pang Y, Repka MX, Tamkins SM, Weise KK; Pediatric Eye Disease Investigator Group. Stereoacuity in children with anisometropic amblyopia. J AAPOS. 2011 Oct;15(5):455-61. doi: 10.1016/j.jaapos.2011.06.007. PMID 22108357
- [Derived] Repka M, Simons K, Kraker R; Pediatric Eye Disease Investigator Group. Laterality of amblyopia. Am J Ophthalmol. 2010 Aug;150(2):270-4. doi: 10.1016/j.ajo.2010.01.040. Epub 2010 May 8. PMID 20451898